CLINICAL TRIAL: NCT04385056
Title: An Open-label, Dose-escalation Study to Evaluate the Use of Umbilical Cord-derived Allogeneic Mesenchymal Stem Cells (UC-MSCs) for the Treatment of Bradykinesia
Brief Title: Evaluate Umbilical Cord-derived Allogeneic Mesenchymal Stem Cells for the Treatment of Bradykinesia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IMAC Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMAC-001
Record Dates: First submitted 2020-05-05; First posted 2020-05-12 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Bradykinesia
MeSH Terms: conditions — Hypokinesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low Dose MSCTC-0010 (Experimental): Participants will receive low-dose cell administration
  Interventions: Biological: MSCTC-0010
- Medium Dose MSCTC-0010 (Experimental): Participants will receive medium-dose cell administration
  Interventions: Biological: MSCTC-0010
- High Dose MSCTC-0010 (Experimental): Participants will receive high-dose cell administration
  Interventions: Biological: MSCTC-0010

INTERVENTIONS:
Biological: MSCTC-0010 — MSCTC-0010 is a suspension product for infusion. The active ingredient is the umbilical cord-derived allogeneic mesenchymal stem cells (US-MSCs).

SUMMARY:
Investigate the safety and tolerability of umbilical cord-derived allogeneic mesenchymal stem cells to treat patients with Bradykinesia.

DETAILED DESCRIPTION:
While the pathophysiological changes that result in the symptoms of bradykinesia are poorly understood, an inflammatory component appears to be involved. Human umbilical cord-derived allogeneic mesenchymal stem cells have documented anti-inflammatory properties, which suggest these cells may be effective at treating Bradykinesia. It is understood that perinatal products are potent immune modulators. It is believed that the positive symptomatic effects are secondary to the modulation of the immune system, and specifically the reduction in pathological inflammation. The study is designed to evaluate the safety and tolerability of umbilical cord-derived allogeneic mesenchymal stem cells to treat patients with Bradykinesia.

ELIGIBILITY:
Inclusion Criteria:

* Age of 55 years or older
* Clinically diagnosed with Parkinsonism
* All subjects, or their authorized representatives, must be adequately informed and understand the nature and risks of the study and must be able to provide a signature and date in the Informed Consent Form (ICF).
* Clinically diagnosed bradykinesia for at least 3 months prior to baseline visit.
* On stable treatment regimen with L-dopa and other anti-parkinsonian treatment for 4 weeks prior to baseline.
* Women of child-bearing potential must undergo a negative serum pregnancy test at the screening assessment.
* Subjects, or their representatives, must be able to communicate effectively with the study staff.
* Subjects, or their authorized representatives, must certify that they are able and willing to follow all protocol requirements and study restrictions.

Exclusion Criteria:

* Subjects who are intolerant of, or unwilling to, participate in all procedures required of this protocol.
* Subjects who cannot tolerate a venipuncture and/or have adequate venous access.
* Inability to ambulate 100 feet independently with or without an assistive device.
* Subjects who have a history of allergy, hypersensitivity, or intolerance to any medications, components, or excipients of the investigational product or procedures, and which cannot be resolved by the staff conducting the study.
* Subjects with a known diagnosis of Atypical Parkinsonian Syndrome e.g.:

  1. Dementia with Lewy Bodies;
  2. Progressive Supranuclear Palsy;
  3. Corticobasal Degeneration;
  4. Multiple System Atrophy;
  5. Other Neurodengerative Conditions.
* Head trauma related to the onset of bradykinesia symptoms.
* History of repeated head injury, hydrocephalus, encephalitis, or cerebral tumors.
* Choreoathetosis
* Any documented abnormality in the brain by CT or MRI, which might contribute to the motor function, e.g., stroke, tumor, or other space-occupying lesions, hydrocephalus, or encephalomalacia.
* Known history of serum or plasma progranulin level < 110.9 ng/mL.
* Disease associated mutation in TDP-34, PGRN, CHMPB2, or VCP genes or any other FTLD Causative genes.
* Intracranial operation, e.g., pallidotomy, thalamotomy, and/or deep brain stiumulation surgery.
* Other known neurodegenerative diseases not underlying the bradykinesia, e.g., Spinocerellar Atropy (SCA), Wilson's Disease, or Amyotrphic Lateral Sclerosis (ALS).
* History of other significant neurological or physciatric disorders including, but not limited to, Alzheimer's disease, Lewy Body Dementia, Prior Disease, stroke, or seizure disorder.
* Psychiatric illness that is unrelated to the Bradykinesia, e.g., severe bipolar or unipolar depression.
* History of neurotoxin exposure.
* History of REM behavior disorder.
* Patients with Hepatocellular Carcinoma (HCC).
* Acute liver failure or episode of hepatic encephalopthy.
* Systolic blood pressure greater than 180 or less than 90 mmHg.
* Diastolic blood pressure greater than 105 or less than 50 mmHg.
* Presence of QTcprolongation or ECG abnormal at screening and judged to be clinically significate by the site investigator.
* Clinically significant cardiovascular disease, e.g., cardiac surgery or myocardial infarction within the last 6 months, unstable angina, congestive heart failure, significant cardaic arrthymia; or cogenitial heart disease.
* Early, symptomatic autonomic dysfunction.
* Any malignancy (other than non-metasticic basal cell carcinoma of the skin) with 5 years of screening.
* Clinically significant lab abnormalities at screening, including creatinine ≥ 2.5 mg/dL, vitam B12 below laboratory normal reference range, or TSH above laboratory normal reference range.
* Current clinically significant hematological, endocrine, cardiovascular, renal, heapatic, gastrointestinal, or neurological disease. For the non-cancerconditions, if the condition has been stable for at least the past year and is judged by the site investigator not to interfere with the patient's participation in the study, the patient may be included.
* A history of alcohol or substance abuse within 1 year prior to screening and deemed to be clinically significant by the site investigator.
* An employee or relative of an employee.
* Subjects who have donated plasma or platelets or had a significant loss of whole blood (480 ml or more) within 30 days.
* Subjects who have received blood or blood products within 30 days prior to screening.
* Treatment with any investigational drugs or device or participation in an investigational drug study within 60 days of screening.
* Women of childbearing potential who are not using at least two forms of medically recognized contraception.
* Female subjects who are pregnant, expecting to become pregnant, or lactating/nursing.
* Any subjects who have a clinically significant abnormal laboratory value.
* Subjects who have been treated with another research product 30 days prior to the screening assessment, or plant to participate in another clinical trial, while in this study. If more than 30 days have passed since participation in another clinical trial, the study staff must ensure that the subject has recovered from any adverse events associated with the research product used.
* Subjects who have a history of any other clinically significant disease or disorder that in the opinion of the Principal Investigator, may place the subject at risk due to participation in the study, or may influence the results of the study.

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-12-15 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Serious Adverse Events and Adverse Events | 12 months
  Number of serious adverse events and adverse events for the duration of the study.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - IMAC Regeneration Center, Paducah, Kentucky
  - Ozzie Smith IMAC Regeneration Center, Chesterfield, Missouri
  - David Price IMAC Regeneration Center, Brentwood, Tennessee

IPD SHARING:
Plan to Share IPD: No